CLINICAL TRIAL: NCT05907473
Title: The Effect of Virtual Reality Therapy Applied in Addition to Conventional Balance Training on Balance and Knee Control in Stroke Patients
Brief Title: The Effect of Virtual Reality Therapy on Balance and Knee Control in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Suleyman Korkusuz, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-77
Record Dates: First submitted 2023-05-24; First posted 2023-06-18 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Chronic Stroke
Keywords: Virtual Reality; Stroke; Knee Hyperextension; Gait Analysis; Activities of Daily Living; Balance
MeSH Terms: conditions — Stroke | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Rehabilitation Group (Experimental): In the conventional rehabilitation program, bed exercises, mat activities, balance exercises inside or outside the parallel bar and walking training will be given to the patients every weekday.
  Interventions: Other: Conventional Rehabilitation
- Virtual Reality Therapy Group (Experimental): The patients in this group will be able to play balance-based games with the Virtual Reality System for 20 minutes, 3 days a week, together with the conventional rehabilitation program.
  Interventions: Other: Virtual Reality Therapy; Other: Conventional Rehabilitation

INTERVENTIONS:
Other: Virtual Reality Therapy — Patients in this group will play balance-based games with the Virtual Reality System.
  Arms: Virtual Reality Therapy Group
Other: Conventional Rehabilitation — In the conventional rehabilitation program, bed exercises, mat activities, balance exercises inside or outside the parallel bar and walking training will be given to the patients every weekday.

SUMMARY:
The aim of study is to determine whether the Virtual Reality training applied in addition to the exercises given inside and outside the parallel bar is effective on balance, daily living activities and knee control in stroke patients.

The hypotheses of the study are:

Hypothesis 1:

H0: Virtual reality training has no effect on balance in stroke patients. H1: Virtual reality training has an effect on balance in stroke patients.

Hypothesis 2; H0: Virtual reality training has no effect on activities of daily living in stroke patients.

H1: Virtual reality training has an effect on daily living activities in stroke patients.

Hypothesis 3; H0: Virtual reality training has no effect on knee control in stroke patients. H1: Virtual reality training has an effect on knee control in stroke patients

DETAILED DESCRIPTION:
In recent years, virtual reality systems are widely preferred technology-assisted rehabilitation methods due to the many advantages they provide in stroke rehabilitation. Virtual reality increases the quality of movement and functional capacity both by providing a sensory environment and by motor learning.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-70
* Having a stroke for the first time
* Patients who can stand and walk independently

Exclusion Criteria:

* Having neglect syndrome
* Being bilaterally affected
* Botulinum toxin application in the last three months
* Having additional neurological diseases such as Parkinson's, multiple sclerosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Computerized Gait Assessment System (Zebris Rehawalk) | Baseline
  Participants will walk at a comfortable walking speed on the treadmill. During the walk, the walk will be recorded with the video camera system integrated into the device. With the help of the system, the knee hyperextension angle during walking will be calculated with the markers placed on the recorded video.
Computerized Gait Assessment System (Zebris Rehawalk) | 6.week (at the end of the training)
  Participants will walk at a comfortable walking speed on the treadmill. During the walk, the walk will be recorded with the video camera system integrated into the device. With the help of the system, the knee hyperextension angle during walking will be calculated with the markers placed on the recorded video.
Barthel Index | Baseline
  This scale consists of 10 items that evaluate nutrition, bathing, self-care, dressing, defecation control, urine control, going to the toilet, ability to move from bed to wheelchair, mobility status such as walking or being dependent on a wheelchair, and stair climbing functions.
Barthel Index | 6.week (at the end of the training)
  This scale consists of 10 items that evaluate nutrition, bathing, self-care, dressing, defecation control, urine control, going to the toilet, ability to move from bed to wheelchair, mobility status such as walking or being dependent on a wheelchair, and stair climbing functions.
Functional Reach Test | Baseline
  It is based on the principle of lifting the arm 90° upwards and reaching forward as far as possible while keeping the feet on the ground. 15 cm. and the risk of falling below 15 cm increases significantly, between 15 and 25 cm. indicates a moderate risk of falling. Values less than 25.4 cm indicate an increased risk of falling.
Functional Reach Test | 6.week (at the end of the training)
  It is based on the principle of lifting the arm 90° upwards and reaching forward as far as possible while keeping the feet on the ground. 15 cm. and the risk of falling below 15 cm increases significantly, between 15 and 25 cm. indicates a moderate risk of falling. Values less than 25.4 cm indicate an increased risk of falling.
Timed Up and Go Test | Baseline
  It is an objective, reliable and simple measure for assessing balance and functional mobility. It can also be used for assessment of fall risk.
Timed Up and Go Test | 6.week (at the end of the training)
  It is an objective, reliable and simple measure for assessing balance and functional mobility. It can also be used for assessment of fall risk.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Yürük, Prof.Dr., Study Chair — Baskent University; Süleyman Korkusuz, MSc, Principal Investigator — Atılım University; Gülşen Taşkın, Assist.Prof, Study Chair — Afyonkarahisar Sağlık Bilimleri University; Melike Sümeyye Cengiz, MSc, Study Chair — Bandırma Onyedi Eylül University; Büşra Seçkinoğulları, MSc, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palacios-Navarro G, Garcia-Magarino I, Ramos-Lorente P. A Kinect-Based System for Lower Limb Rehabilitation in Parkinson's Disease Patients: a Pilot Study. J Med Syst. 2015 Sep;39(9):103. doi: 10.1007/s10916-015-0289-0. Epub 2015 Aug 12. PMID 26265237
- [Background] Park DS, Lee DG, Lee K, Lee G. Effects of Virtual Reality Training using Xbox Kinect on Motor Function in Stroke Survivors: A Preliminary Study. J Stroke Cerebrovasc Dis. 2017 Oct;26(10):2313-2319. doi: 10.1016/j.jstrokecerebrovasdis.2017.05.019. Epub 2017 Jun 9. PMID 28606661
- [Derived] Korkusuz S, Taskin G, Korkusuz BS, Ozen MS, Yuruk ZO. Examining the effects of non-immersive virtual reality game-based training on knee hyperextension control and balance in chronic stroke patients: a single-blind randomized controlled study. Neurol Sci. 2025 Mar;46(3):1267-1275. doi: 10.1007/s10072-024-07830-z. Epub 2024 Oct 28. PMID 39466327